CLINICAL TRIAL: NCT02046759
Title: A Comparative Study of an Integrated Pharmaceutical Care Plan and a Routine Care in Bronchial Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rana Rasheed Ibrahim Farrag, Pharmacist, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Asthma-001
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pharmacist-Intervention (Experimental)
  Interventions: Other: Pharmacist- Intervention
- Routine Care (Active Comparator)
  Interventions: Other: Routine Care

INTERVENTIONS:
Other: Pharmacist- Intervention — Patients received additional education on basic facts about asthma, role of medications, the difference between long-term control medications and quick-relief medications, as well as patient skills in the first visit then reinforcement every two weeks.. The importance of proper inhaler technique, avoidance of asthma triggers and self-monitoring of asthma were also highlighted. Visual aids, physical demonstration as well as written information resources were supplied. Asthma care plans were tailored to patient needs and preferences. Patients were informed how to detect early signs of worsening asthma, when and how to seek medical care as appropriate.
  Other Names: Patient Education; Asthma Action Plan; Shared Decision Making
  Arms: Pharmacist-Intervention
Other: Routine Care — Patients received usual care delivered by physician without pharmacist intervention. Patients were prescribed asthma medication with summarized basic information on asthma and medication use. Follow-up visits were not planned on consistent basis, but rather individually according to the disease status. No asthma action plans were provided.
  Arms: Routine Care

SUMMARY:
The aim of the study is to compare the effect of asthma care by clinical pharmacist intervention versus routine care on asthma control.

ELIGIBILITY:
Inclusion Criteria:

* patient with clinical diagnosis of bronchial asthma
* responsible for administering their own asthma medications.

Exclusion Criteria:

* patients who were not responsible for administering their own asthma medications.
* patients with cognitive defects, other pulmonary disease e.g. Chronic Obstructive Pulmonary Disease (COPD), experiencing illness with asthma-like symptoms e.g. Congestive Heart Failure, evidence of fixed airway obstruction
* patients unavailable for 2-month follow-up.
* patients who did not provide written informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Asthma Control Questionnaire | at baseline & after 2 months of therapy

SECONDARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1%) | at baseline & after 2 months of therapy
Rescue Medication SABA (number of puffs used most days) | at baseline & after 2 months of therapy
Inhaled Corticosteroid Use (number of puffs used/day) | at baseline & after 2 months of therapy
Number of courses of systemic steroid used | During 2 months of therapy
Number of ER visits/ Hospitalization | During 2 months of therapy

OTHER OUTCOMES:
Assessment of Inhalation Technique | at baseline and after 2 months of therapy
Patient Adherence to Therapy | 2 months of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Rana R Farrag, Principal Investigator — Ahram Canadian University
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt